CLINICAL TRIAL: NCT07100886
Title: Long-Term Safety and Efficacy Evaluation of Seal-G and Seal-G MIST Surgical Sealants for Anastomosis Protection in Colon Surgery [PMCF Study Continuation]
Brief Title: Seal-G/ Seal-G MIST Long-Term Follow-up PMCF (Continue) Study
Status: Not yet recruiting | Type: Observational
Sponsor: Advanced Medical Solutions Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: DLG-072-13
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Colon Anastomosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective Treatment Group: Patients who underwent colectomy and anastomosis coverage with Seal-G / Seal-G MIST as part of the previous PCMF study protocol (#DLG-072-06)
  Interventions: Other: long-term follow up visit
- Retrospective Control Group: Patients who underwent colon resection with primary anastomosis (SOC) (comparable population)
  Interventions: Other: long-term follow up visit

INTERVENTIONS:
Other: long-term follow up visit — Phone call questionnaire- retrospective treatment arm Phone call questionnaire- retrospective control arm

SUMMARY:
Postoperative complications following colon anastomosis surgery, such as adhesions, stenosis, stricture and obstruction, can significantly impact patient outcomes. The use of surgical sealants has been proposed as a means to mitigate anastomotic complications by providing a protective barrier over the anastomosis site, reducing the risk or the severity of anastomotic leak. The previous post-market clinical follow-up (PMCF) study assessed the short-term safety and performance of SEAL-G surgical sealants in preventing anastomotic leaks and early post-operative complications. However, long-term data are needed to establish its sustained safety and effectiveness.

This continuation study aims to evaluate the long-term impact of the SEAL-G/MIST surgical sealant on post-operative complications over 12+ months after surgery. The study will compare complication rates in patients treated with the surgical sealant to a retrospective comparable control group who underwent similar procedures without the sealant.

DETAILED DESCRIPTION:
The study is designed as an observational, retrospective-controlled, long-term follow-up, multi-center post-market clinical follow-up (PMCF) study.

For the Retrospective Treatment Group, 3 out of the 8 sites participated in the previous PMCF study (#DLG-072-06), will be included with a total of 104 patients who received the Seal-G / Seal-G MIST surgical sealant during colon anastomosis surgery 2-4 years ago (during 2021-2023). The following sites were selected due to relatively large number of participants in the previous study and according to their ability to comply with the current study procedures.

For the Retrospective Control group, screening will be performed at each site, for a matching number of subjects from a comparable population (i.e age; BMI; surgery procedure (2-4 years ago); etc.) that did not receive the sealant treatment. Phone Questionnaire: Long-term follow-up visit should be performed via Phone call Questionnaire. Patients will be contacted (including Oral informed consent) to assess long-term outcomes relating to the colon anastomosis surgery they underwent 2-4 years ago.

* Incidence of adhesions, stenosis, and obstruction (reported during the Physician questionnaire and confirmed by medical records review where possible).
* Need for reoperation due to complications.
* Use of additional treatments relating to anastomosis complications (e.g., anti-adhesion therapy, bowel obstruction management).

ELIGIBILITY:
Inclusion Criteria:

* Treatment Group: Patients participated and completed all visits in the previous PMCF study (treatment group; #DLG-072-06)
* Control Group: comparable retrospective subjects that meet the same inclusion criteria specified in #DLG-072-06.
* Both Treatment & Control group:

Willing to comply with long-term follow-up assessment (including oral consent).

Exclusion Criteria:

* Both Treatment & Control group:

Patients who are unable or unwilling to complete the phone questionnaire.

- Control group: Subjects that would have been excluded according to the previous PMCF study #DLG-072-06 exclusion criteria.

* Patients with missing or incomplete medical records that prevent retrospective comparison.
* Patients that during the original surgery received any treatment on the anastomosis (sealant/glue) except for the anastomosis closure technique (sutures/staple).
* Original surgery included stoma creation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For the Retrospective Treatment Group, 3 out of the 8 sites participated in the previous PMCF study (#DLG-072-06), will be included with a total of 104 patients who received the Seal-G / Seal-G MIST surgical sealant during colon anastomosis surgery 2-4 years ago (during 2021-2023). The following sites were selected due to relatively large number of participants in the previous study and according to their ability to comply with the current study procedures.
  For the Retrospective Control group, screening will be performed at each site, for a matching number of subjects from a comparable population (i.e age; BMI; surgery procedure (2-4 years ago); etc.) that did not receive the sealant treatment.
Sampling Method: Non-Probability Sample
Enrollment: 208 (Estimated)
Dates: Start 2025-08-04 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Rate of reoperation due to anastomotic complications | 1 year post-surgery
Assessment of long-term anastomotic complications (i.e. adhesions, stenosis, stricture, and obstruction) | 1 year post-surgery
  At least one complication within the 1 year interval

SECONDARY OUTCOMES:
The incidence of anastomotic complications (i.e. adhesions, stenosis, stricture, and obstruction) | 1-4 years post-surgery
The incidence of hospitalization due to anastomotic complications | 1-4 years post-surgery
The incidence of reoperation due to anastomotic complications | 1-4 years post surgery
The incidence of anastomotic leaks (Clinical/sub-clinical) | 30 day post surgery

IPD SHARING:
Plan to Share IPD: Undecided